CLINICAL TRIAL: NCT03700177
Title: Ropivacaine 0,2% Plus Dexamethasone Versus Ropivacaine 0,2% Plus Placebo in Modified Pectoral Block - a Randomized, Double-blind, Prospective Trial
Brief Title: Ropivacaine 0,2% Plus Dexamethasone Versus Ropivacaine 0,2% Plus Placebo in Modified Pectoral Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Effect of Drugs; Breast Pain; Anesthesia, Local
MeSH Terms: conditions — Mastodynia | interventions — Dexamethasone; Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ropivacaine + dexamethasone (Active Comparator): Every participant receives general anesthesia and a modified pectoral nerve block for breast surgery. Participants of this arm receive single-shot ropivacaine (0,2%, 30ml) plus 2ml dexamethasone (8mg).
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine Injection [Naropin]
- ropivacaine + placebo (Placebo Comparator): Every participant receives general anesthesia and a modified pectoral nerve block for breast surgery. Participants of this arm receive single-shot ropivacaine (0,2%, 30ml) plus 2ml placebo (NaCl 0,9%).
  Interventions: Drug: Placebo; Drug: Ropivacaine Injection [Naropin]

INTERVENTIONS:
Drug: Dexamethasone — modified pectoralis block for breast surgery with ropivacaine combined with dexamethasone 8mg.
  Other Names: Dexabene
  Arms: ropivacaine + dexamethasone
Drug: Placebo — modified pectoralis block for breast surgery with ropivacaine combined with placebo (NaCl 0,9%).
  Other Names: sodium chloride (NaCl) 0,9%
  Arms: ropivacaine + placebo
Drug: Ropivacaine Injection [Naropin] — 30ml (=60mg) for modified pectoralis block (thoracic regional fascial plane block)
  Other Names: Naropin

SUMMARY:
To find out if dexamethasone used as adjuvant to ropivacaine, a long-lasting local anesthetic, prolongs the duration of modified pectoral nerve block in women undergoing breast surgery.

DETAILED DESCRIPTION:
Breast surgeries are one of the most common forms of surgery conducted in hospitals, and even relatively minor interventions can be associated with significant postoperative pain. The most common surgical procedure for breast cancer is modified radical mastectomy, which means removing a generous amount of skin and the entire breast with axillary evacuation. According to the literature, up to 50% of breast surgery patients experience severe acute postoperative pain, with 10-40% breast cancer patients experiencing pain a year or more after surgery.

Poorly controlled postoperative pain has negative physiological and psychological consequences. Furthermore, effective acute pain control preserves immune function both by suppressing surgical stress response and decreasing the need for general anesthetics and opioids in the perioperative period.

The ultrasound-guided modified, pectoral nerve block is a frequently used, easy, and reliable technique to provide complete analgesia during and after breast surgery. A major limitation to its use for postoperative analgesia is that the analgesic effect lasts only a few hours, after which moderate to severe pain at the surgical site may result in the need for alternative analgesic therapy. Several adjuvants have been used to prolong the analgesic duration of peripheral nerve block, including perineural/interfascial or intravenous dexamethasone.

Our aim is to explore the efficacy of 8 mg dexamethasone added to US-guided modified pectoral nerve block on postoperative pain in patients undergoing major breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* a American Society of Anesthesiologists (ASA) score of 1 or 2
* weight: body mass index (BMI) 18 - 35 kg/m2
* informed consent
* elective, unilaterale breast surgery

Exclusion Criteria:

* bleeding disorders
* any known allergy to the medication
* diabetes mellitus
* any disease that leads to alterations in the corticosteroid physiology
* drug-dependency
* BMI <18 or > 35
* systemic infections
* psychiatric diseases, that are associated with an alteration in the perception of pain
* tumor spread at the site of injection
* inflammation at the site of injection
* pregnancy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
morphine consumption in the first 72 hours | 72 hours
  every participants receives a morphine pump (PCA) to exactly measure opioid-consumption

SECONDARY OUTCOMES:
VAS-scores in the first 72 hours | 72 hours
  Every participant is being repeatedly asked to score pain intensity on the visual-analog scale (VAS). This is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points (0-10). VAS is the most common scale for pain quantification worldwide. A VAS-scale of 0 indicates "no pain" and 10 indicates "worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Karl Lindner, Prof.Dr., Study Director — Department of Anesthesia and Intensive Care
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No